CLINICAL TRIAL: NCT07189325
Title: A Prospective Randomized Non-inferiority Trial Comparing Anti-CD20 Maintenance Versus De-Escalation Strategy In Relapsing-Remitting Multiple Sclerosis
Acronym: DESIRE MS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECHMPL23_0397; 2024-513292-40-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-23; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Relapsing-Remitting Multiple Sclerosis (RRMS); Anti-CD20 Therapy
Keywords: Multiple Sclerosis; High efficacy therapies; de-escalation; adverse events; relapses; escalation
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Recurrence | interventions — Dimethyl Fumarate; teriflunomide; Glatiramer Acetate; Interferon-beta; ocrelizumab; Rituximab; ofatumumab

STUDY DESIGN:
Intervention Model Description: Multi-center, prospective, comparative, randomized into two parallel (1:1) arms, open to treatment with blinded endpoint (PROBE) non-inferiority trial comparing, over 3 years, the maintenance of anti-CD20 therapies and a de-escalation strategy:
  * Experimental group: Patients randomized in the experimental group will be treated with platform therapies (Dimethyl Fumarate, Diroximel fumarate, Teriflunomide, Glatiramer Acetate, Beta-interferons) according to treatments' authorization from the day of randomization to M36.
  * Control group: Patients randomized in the control group will be treated every 6 months (or, up to one year, at the same interval dosing) for patients with anti-CD20 (ocrelizumab, rituximab) or every 4 weeks for patients with subcutaneous anti-CD20 (ofatumumab) from the day of randomization to M36.
  In both groups, each patient will have a treating neurologist and a blinded examinator who will perform blinded EDSS evaluations and assessment of suspected relapses.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Patients randomized in the experimental group will be treated with platform therapies (Dimethyl Fumarate, Diroximel fumarate, Teriflunomide, Glatiramer Acetate, Beta-interferons) according to treatments' authorization from the day of randomization to M36.
  Interventions: Drug: Platform therapies (Dimethyl Fumarate, Teriflunomide, Glatiramer Acetate, Beta-interferons)
- Control Group (Active Comparator): Patients randomized in the control group will be treated every 6 months (or, up to one year, at the same interval dosing) for patients with anti-CD20 (ocrelizumab, rituximab) or every 4 weeks for patients with subcutaneous anti-CD20 (ofatumumab) from the day of randomization to M36.
  Interventions: Drug: Anti-CD20 therapies (Ocrelizumab, Rituximab, Ofatumumab)

INTERVENTIONS:
Drug: Platform therapies (Dimethyl Fumarate, Teriflunomide, Glatiramer Acetate, Beta-interferons) — Patients randomized in the experimental group will be treated with platform therapies (Dimethyl Fumarate, Diroximel Fumarate, Teriflunomide, Glatiramer Acetate, Beta-interferons) according to treatments' authorization from the day of randomization to M36 described below.
  Patients will receive appropriate information and recommendation for the initiation of the chosen platform treatment as mention in the SmPC by treating neurologist or a member of the investigating team. If therapies are not tolerated, a therapeutic switch to other platform therapies will be possible. Any switch to a disease modifying therapy not listed as platform therapy will be considered as a major protocol deviation (see statistics).
  Patients are allowed to switch from any platform DMT to another platform DMT.
  Arms: Experimental Group
Drug: Anti-CD20 therapies (Ocrelizumab, Rituximab, Ofatumumab) — Patients randomized in the control group will be treated every 6 months (or at previous extended interval dosing) for patients with anti-CD20 (Ocrelizumab, Rituximab) or every 4 weeks for patients with subcutaneous anti-CD20 (Ofatumumab) from the day of randomization to M36. If therapies are not tolerated, a therapeutic switch to other anti-CD20 therapy will be possible. Any switch to a disease modifying therapy not listed as anti-CD20 therapy will be considered as major protocol deviation (see statistics).
  Patients are allowed to switch from any anti-CD20 to another anti-CD20.
  Arms: Control Group

SUMMARY:
Multiple sclerosis (MS), the main central nervous system autoimmune disorder, is the first cause of non-traumatic disability in young adults and has thus significant individual consequences with elevated public health cost. It commonly starts during the third and fourth decades. Over the last twenty years, several disease-modifying therapies with variable benefit/risk profiles have been introduced leading to dramatic changes in the prognosis of MS.

First, several moderately effective therapies , with good safety profile, have allowed to decrease the frequency of relapses along with a possible, albeit limited, effect on medium- and long-term disability.

More recently highly effective therapies (HET), with immunosuppressive properties, have dramatically reduced clinical and MRI disease activity and significantly improved patient's prognosis.

Anti-CD20 therapies (B-cells depleting therapies, given either intravenous or subcutaneous), one of the main HET, have demonstrated higher efficacy than platform therapies in several phase 3 randomized clinical trials and their use within the very first years of the disease seems to be associated with improved long-term outcomes.

Taking all of this into account, the investigators hypothesize that RRMS patients who experience a de-escalation from anti-CD20 therapies to platform therapies after 40 years will not experience disease activity accrual and disability worsening.

ELIGIBILITY:
Inclusion criteria :

* Patients ≥40 years at inclusion
* Patients with relapsing remitting multiple sclerosis at inclusion (according to 2017 McDonald criteria) treated with anti-CD20 for at least the last 3 years. For patients treated with IV ocrelizumab or rituximab at extended interval dosing, a maximum interval of 12 months between perfusions during the year before inclusion visit is required.
* No evidence of disease activity for the last 3 years on anti-CD20 (No relapse AND no new/enlarged MRI lesion)
* Brain MRI performed according to OFSEP protocol within a maximum of 6 months before randomization

Non-inclusion criteria :

* Secondary or primary progressive MS at inclusion
* Previous experience of treatment failure in patients treated with natalizumab, fingolimod, rituximab, ocrelizumab, mitoxantrone, alemtuzumab or cladribine
* Treatment with high dose corticosteroids during the 30 days preceding inclusion
* Contraindication to MRI
* Severely immunocompromised state
* Current severe active infection
* Known active malignancy
* Severe heart failure (New York Heart Association Class IV) or severe, uncontrolled cardiac disease
* Severe hepatic impairment (Child-Pugh class C)
* Significantly impaired bone marrow function or significant anaemia, leukopenia, neutropenia or thrombocytopenia
* Severe renal impairment undergoing dialysis
* Severe hypoproteinaemia, e.g. in nephrotic syndrome
* Current severe depression and/or suicidal ideation
* Suspected or confirmed progressive multifocal leukoencephalopathy (PML)
* Any condition that, in the opinion of the investigator, would interfere with the interpretation of patient safety or place the patient at high risk for treatment-related complications
* Participation in another therapeutic trial in the last 6 months
* Protected population according to articles of the French Public Health Code (e.g. patients under law protection, prisoners, pregnant, parturient or lactating women, and patients under guardianship/curatorship)
* All women of childbearing age not using effective contraception during the study
* Subjects not covered by public health insurance
* Failure to obtain written informed consent after a reflection period

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Relapse | From Day 0 to Month 36
  Presence of at least one clinical relapse defined as new or worsening symptoms related to MS resulting in objective signs on neurological examination in the absence of any potential trigger not related to MS.
New/enlarged MRI lesions | From Day 0 to Month 36
  New/enlarged T2/FLAIR lesion on MRI scans to assess MRI disease activity .

SECONDARY OUTCOMES:
Relapse | From Day 0 to Month 36
  Presence of at least one clinical relapse defined as new or worsening symptoms related to MS resulting in objective signs on neurological examination in the absence of any potential trigger not related to MS
Expanded Disability Status Scale (EDSS) | From Day 0 to Month 36
  EDSS to compare disability between both groups. This score is expressed from 0 (no disability) to 10 (multiple sclerosis-related death) and incorporates evaluation of the following neurological systems (pyramidal, sensory, cerebellar, sphincter, cognitive, and cranial pairs)
Brain MRI (T2/FLAIR Lesions) | From Day 0 to Month 36
  MRI scans to compare new/enlarged T2/FLAIR lesions between both groups.
Number of adverse events and severe adverse events | From Day 0 to Month 36
  To compare adverse events and severe adverse events between both groups.
Number of infections and serious infections | From Day 0 to Month 36
  To compare infections and serious infections between both groups.
B-cell count (CD19/CD20 B cells) | From Day 0 to Month 36
  B-cell count (CD19/CD20 B cells) to compare C• B-cells repopulation (CD19/CD20+ B-cells) between both groups.
Serum immunoglobulin (IgG, IgA, IgM) levels | From Day 0 to Month 36
  Serum immunoglobulin (IgG, IgA, IgM) levels to compare • Immunoglobulin (IgG, A, M) levels changes between both groups.

OTHER OUTCOMES:
Multiple Sclerosis Functional Composite (MSFC) | From Day 0 to Month 36
  MSFC including the 9-Hole Peg Test (9HPT), Timed 25 Foot Walk (T25FW), and Paced Auditory Serial Addition Test (PASAT) to compare functional disability between both groups.
The Computerised Speed Cognitive Test (CSCT) | From Day 0 to Month 36
  CSCT a cognitive test to compare the detection of information speed disorders between both groups.
Neurofilament Light Chains (sNfL) Serum Concentration | From Day 0 to Month 36
  Neurofilament Light Chains (sNfL) Serum Concentration to compare change of serum Neurofilament light chains bteween both groups.
The 5 Level European Quality of Life 5 Dimensions (EQ5D-5L) | From Day 0 to Month 36
  EQ5D-5L questionnaire to compare the generic quality of life between both groups.
MUSICARE | From Day 0 to Month 36
  MUSICARE, self-report questionnaire to compare the experience of both patients and caregivers of quality of care in MS between both groups.
CD27+ memory B-cell count | From Day 0 to Month 36
  CD27+ memory B-cell count to compare CD27+ memory B-cells repopulation between both groups.
Patient-level cost | From Day 0 to Month 36
  Healthcare consumption collected via data from the SNDS (French Health Insurance Database) to assess medico-economic impact.

CONTACTS AND LOCATIONS:
Locations (1):
- Neurology Department, Hospital Gui de Chauliac, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided